CLINICAL TRIAL: NCT00119197
Title: Safety and Immunogenicity of a Killed, Oral Cholera Vaccine in Indian Subjects in Eastern Kolkata, West Bengal
Brief Title: Safety and Immunogenicity of Oral Cholera Vaccine in Kolkata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Indian Council of Medical Research (Other Government); Shantha Biotechnics Limited (Industry)
Responsible Party: Director General, International Vaccine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-8-ph2
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Cholera
Keywords: watery diarrhea; cholera vaccine
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Killed Whole Cell Oral Cholera Vaccine
  Interventions: Biological: killed whole cell oral cholera vaccine
- 2 (Placebo Comparator): Heat-killed E. coli
  Interventions: Biological: Heat Killed E. coli

INTERVENTIONS:
Biological: killed whole cell oral cholera vaccine — Bivalent oral killed cholera vaccine: each dose of this vaccine contains:
  * Inactivated V.Cholerae Inaba (569B), Classical biotype - 25.109 cells
  * Inactivated V.Cholerae Ogawa (Cairo 50) Classical biotype - 25.109 cells
  * Inactivated V.Cholerae Inaba (Phil 6973) El Tor biotype - 50.109 cells
  * Inactivated V.Cholerae O139 - 50.109 cells
  each 1.5 mL dose given orally, two doses given 14 days apart
  Arms: 1
Biological: Heat Killed E. coli — Escherichia coli K12 strain placebo: each dose of placebo contains heat-killed E. coli K12 strain in an amount whose optical turbidity is identical to that for the cholera vaccine.
  Each 1.5 mL dose given orally, two doses given 14 days apart
  Arms: 2

SUMMARY:
The purpose of the study is to confirm the safety and immunogenicity of the oral killed bivalent cholera vaccine in adult and pediatric volunteers in Eastern Kolkata, West Bengal, India.

DETAILED DESCRIPTION:
Cholera remains to be a serious public health problem worldwide. In the mid-1980s following technology transfer from Sweden, Vietnamese scientists developed and produced an oral killed monovalent cholera vaccine for Vietnam's public health programs. A 2-dose regimen of this vaccine has been shown to be safe and efficacious. Subsequently, a bivalent vaccine was developed containing the newly emergent O139 V. cholerae. This vaccine has several advantages over the existing Swedish vaccine. It confers protection against the El Tor biotype in younger children, is considerably less expensive, does not require a buffer during administration and does not require strict cold chain requirements. However, this vaccine is not licensed for use in countries other than Vietnam.

Through IVI, an agreement between VABIOTECH in Hanoi and Shantha Biotechnics PVT, LTD in India has been reached that will make the bivalent vaccine available in India. A double-blind randomized phase III trial in a cholera-endemic area would be necessary to demonstrate the efficacy of this vaccine in other settings. This would pave the way for the introduction of the vaccine into the national immunization programme in India and the internationalization of this vaccine and licensure in other countries where it is needed. Prior to the phase III trial, a phase II study will be performed among adults and children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant adults aged 18-40 years and children aged 1-17 years

Exclusion Criteria:

* Diarrhea during the past week
* Antibiotic and anti-diarrheal medicine use during the past week
* One or more episodes of diarrhea or abdominal pain lasting for 2 weeks during the past 6 months
* Abdominal pain, nausea, vomiting, loss of appetite or generalized ill feeling for the past 24 hours
* Pregnancy

Ages: 12 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2005-08; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
adverse events | immediate events - 30 minutes after each dose, adverse events - for 3 days following dose, serious adverse events throughout study - 28 days

SECONDARY OUTCOMES:
serum vibriocidal antibody response | baseline and 14 days after second dose

CONTACTS AND LOCATIONS:
Overall Officials: Sujit K Bhatttacharya, MD, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India

REFERENCES:
- [Background] Mahalanabis D, Lopez AL, Sur D, Deen J, Manna B, Kanungo S, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Rao R, Holmgren J, Clemens J, Bhattacharya SK. A randomized, placebo-controlled trial of the bivalent killed, whole-cell, oral cholera vaccine in adults and children in a cholera endemic area in Kolkata, India. PLoS One. 2008 Jun 4;3(6):e2323. doi: 10.1371/journal.pone.0002323. PMID 18523643